## Effect of Modulating CYP3A4 Activity on Mineral Homeostasis NCT02019875 06/16/2016

We summarized demographic characteristics by treatment group using mean (SD) for continuous variables and frequency (percent) for categorical variables. We defined the baseline value of each analyte to be the average of the three pre-randomization measurements, and the post-treatment value to be the analyte measurement after 14 days of treatment. We then used a linear mixed model with random intercepts and main effects for treatment group, the indicator of time (pre- vs. post-treatment), and the interaction of the two. From this model, we extracted the pre-treatment and post-treatment means, the change in analyte comparing pre- vs post-treatment for each group, and the difference in change in analyte comparing each active treatment group with the change observed in the water group. We used a Wald test to test each difference in change compared with water, and a global Wald test to test the null hypothesis that all pre- vs post-treatment changes were the same across treatment group.